CLINICAL TRIAL: NCT07153055
Title: Phase I/II Trial of Lurbinectedin With Osimertinib in Transformed Small Cell Lung Cancer
Brief Title: Lurbinectedin With Osimertinib in Transformed Small Cell Lung Cancer
Acronym: LOTS
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Misty Shields (Other)
Collaborators: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor-Investigator, Misty Shields, Adjunct Assistant Professor of Medical & Molecular Genetics, Indiana University
Organization: Indiana University (Other)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CTO-IUSCCC-0891
Record Dates: First submitted 2025-08-26; First posted 2025-09-03 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Small Cell Lung Cancer ( SCLC ); Transformed Small Cell Lung Cancer
Keywords: EGFR mutations
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — PM 01183; osimertinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Phase I Does De-Escalation (Experimental): 3.2 mg/m2 or 2.6 mg/m2 dose of lurbinectedin with 80 mg or 40 mg daily dose of osimertinib. This will occur day 1 of each 21 day cycle.
  Interventions: Drug: Lurbinectedin; Drug: Osimertinib
- Phase II Dose Expansion (Experimental): 3.2 mg/m2 or 2.6 mg/m2 dose of lurbinectedin with 80 mg or 40 mg daily dose of osimertinib. This will occur day 1 of each 21 day cycle.
  Interventions: Drug: Lurbinectedin; Drug: Osimertinib

INTERVENTIONS:
Drug: Lurbinectedin — Two lurbinectedin does of 3.2 mg/m2 or 2.6 mg/m2. The initial starting dose is 3.2 mg/m2. Patients will receive lurbinectedin, until disease progression or unacceptable toxicity, once every 21 days.
Drug: Osimertinib — Two osimertinib does of 80 mg or 40 mg orally once daily, as assigned by the dose de-escalation cohort for each 21 day cycle.

SUMMARY:
This open-label, Phase I/II trial is studying the safety and effectiveness of an experimental drug combination, lurbinectedin with osimertinib, against a rare type of cancer known as transformed small cell lung cancer (SCLC).

DETAILED DESCRIPTION:
This is an open label prospective multicenter Phase Ib/II trial utilizing a Bayesian Optimal Interval (BOIN) dose-finding design to identify the maximum tolerated dose (MTD) based on DLTs of lurbinectedin and osimertinib. DLT period is 21 days beginning on C1D1. Once the MTD has been identified, 10 subjects total will be enrolled in a Phase II expansion. This number includes the 3 initial subjects in the corresponding MTD group. Subjects will receive a combination of lurbinectedin every 21 days and osimertinib daily, until progression or unacceptable toxicities.

ELIGIBILITY:
Inclusion Criteria

1. ≥ 18 years old at the time of informed consent.
2. Ability to provide written informed consent and HIPAA authorization.
3. Must have a histologically or cytologically confirmed transformation to small cell lung carcinoma/cancer.
4. Must have an initial diagnosis of EGFR altered (EGFR-mutated) non-small cell lung cancer and received EGFR targeted therapy (TKI) osimertinib, and does not demonstrate evidence of acquired molecular underpinnings (i.e., presence of a MET amplification >6 copies or EGFR C797S) resulting in progression on osimertinib, aside from histologic transformation to small cell lung cancer. Interruptions of osimertinib prior to enrollment on study is permitted.

   Note: Tissue specimens from archival tissue are encouraged but not required for enrollment.
5. Patients who have received platinum (cisplatin or carboplatin)/etoposide after histologic transformation are permitted on study. Receipt of last cycle of therapy should be at least 3 weeks prior to initiation of treatment on study. Last exposure to immunotherapy such as anti-PD-L1 should be at least four weeks from treatment to initiation of treatment on study. Patients who decline to receive platinum/etoposide after SCLC transformation, for personal preferences or considered medical ineligible for this regimen, may be considered for this study, subject to investigator discretion.
6. Must have measurable disease per RECIST (version 1.1).
7. ECOG performance status ≤ 2.
8. Adequate laboratory functions on baseline testing within 21 days of enrollment, as defined as:

   a. Hematologic parameters: i. Absolute neutrophil count (ANC) ≥ 1.5x109/L ii. Platelet count (Plt) ≥ 100x109/L b. Hepatic parameters: i. Total bilirubin ≤ 1.5x upper limit of normal (ULN); for patients with suspected/documented Gilbert's syndrome, total bilirubin ≤ 3x ULN.

   ii. AST ≤ 3x ULN. iii. ALT ≤ 3x ULN. c. Renal parameters: i. Creatinine clearance (CrCl) or estimated glomerular filtration rate (eGFR, calculated per institutional standards) should be > 30 mL/min.
9. Women of childbearing potential must have a negative pregnancy test within 21 days of protocol registration. Women are considered to have childbearing potential (regardless of sexual orientation, having undergone a tubal ligation, or remaining celibate by choice) unless they meet one of the following criteria:

   i. Has achieved menarche at some point; or ii. Has not undergone a hysterectomy or bilateral oophorectomy; or iii. Has not been naturally postmenopausal for at least 12 consecutive months (i.e., has had menses at any time in the preceding 12 consecutive months).
10. Women of childbearing potential and men with any partners of child-bearing potential must agree to use 2 forms of effective contraception throughout the study and for 6 months after the last study treatment.

    Note: Acceptable methods of birth control include abstinence, partner with previous vasectomy, placement of an intrauterine device (IUD), condom with spermicidal foam/gel/film/cream/suppository, diaphragm or cervical vault cap, or hormonal birth control (pills or injections).
11. Male subjects must agree to refrain from donating sperm during the study and for 6 months after the last study treatment. Female subjects must agree to refrain from donating eggs during the study and for 6 months after the last study treatment.

Exclusion Criteria

1. Patients who have tumors harboring EGFR exon 20 insertion alterations, EGFR C797S, or known mechanisms of resistance to osimertinib (i.e., MET amplification) aside from histologic transformation to SCLC.
2. Patients who are pregnant (treatment can cause fetal harm) and/or breastfeeding.
3. Symptomatic or unstable brain metastases, requiring > 2 mg dexamethasone orally daily, or received palliative radiation to the CNS within 2 weeks of enrollment.
4. Patients with known history of interstitial lung disease (ILD) or pneumonitis (> grade 1) or ILD/pneumonitis (> grade 1) related to antineoplastic drug treatment.
5. Prior history of documented Stephen Johnson Syndrome (SJS), toxic epidermal necrolysis (TEN), erythema multiforme major (EMM), or aplastic anemia on osimertinib.
6. History of congenital long QTc syndrome or mean resting QTc >500 msec at screening with two replicated EKGs at baseline screening for the study.
7. History of ongoing unstable or uncontrolled cardiac conditions, including documented cardiomyopathy or symptomatic congestive heart failure (defined as New York Heart Association (NYHA) class III or IV).
8. Prior history of documented severe allergic or anaphylactic reaction to osimertinib.
9. Prior history of documented aplastic anemia with osimertinib.
10. Prior history of documented allergic or anaphylactic reactions to inactive ingredients of lurbinectedin, including sucrose, lactic acid, and sodium hydroxide.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-05 (Estimated); Primary Completion 2029-04 (Estimated); Study Completion 2029-10 (Estimated)

PRIMARY OUTCOMES:
Grade 3 or dose-limiting toxicities | Within 30 days after your last dose of study treatment.
  The number of incidences of grade 3 or dose-limiting toxicities of the combination of lurbinectedin with osimertinib assessed using NCI CTCAE v5.0 criteria.

SECONDARY OUTCOMES:
Progression-free survival | Within 30 days after your last dose of study treatment.
  The average length of time of progression-free survival (PFS) of the combination of lurbinectedin with osimertinib.

CONTACTS AND LOCATIONS:
Overall Officials: Misty D Shields, MD, PhD, Principal Investigator — Indiana University Melvin and Bren Simon Comprehensive Cancer Center
Locations (1):
- Indiana University Melvin and Bren Simon Comprehensive Cancer Center, Indianapolis, Indiana, United States